CLINICAL TRIAL: NCT03132493
Title: A Retrospective, Multicenter and Observational Study of Nivolumab Monotherapy Treatment in Subjects With Advanced or Metastatic Squamous (Sq) or Non-Squamous (Non-Sq) Non-Small Cell Lung Cancer (NSCLC) Who Have Received at Least One Prior Systemic Regimens for the Treatment of Stage IIIb/IV NSCLC Within the Expanded Access Program (EAP) in SPAIN
Brief Title: Nivolumab in the Real World: Analysis of the Expanded Use in Spanish Patient
Acronym: NIVEX
Status: Completed | Type: Observational
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 16/05_NIVEX
Record Dates: First submitted 2017-04-25; First posted 2017-04-27 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML — nivolumab 3 mg/kg as an intravenous infusion every 2 weeks until progression
  Other Names: Opdivo

SUMMARY:
The investigators will be retrospectively review the case note of patients registered in the EAP of Nivolumab.

A standard anonymous data collection form will be used to collect data and to analyze it.

Patients with advanced Non-Small Cell Lung Cancer previously treated and included in the SPANISH expanded access programme of nivolumab.

DETAILED DESCRIPTION:
This study will help to understand the efficacy of Nivolumab in the real world setting within the SPANISH expanded access programme.

The main objective of this study is to evaluate nivolumab efficacy in terms of Overall Survival (OS), Progression Free Survival (PFS), Overall Response Rate (ORR) and safety in the clinical practice.

The efficacy variables will be assessed for patients (squamous vs non-squamous) who received second line therapies or third lines and subsequent lines and also, long responders will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Squamous or Non-Squamous, non small cell lung cancer (NSCLC), Stage IIIb/IV (histologically or cytologically confirmed), relapsed after 1 prior platinum-based systemic treatment and who received treatment within the SPANISH expanded access programme of nivolumab (EAP)
2. Alive patients must have signed and dated an IRB/IEC-approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care

Exclusion Criteria:

1. Alive patients who do not want to sign and date an IRB/IEC-approved written informed consent form
2. Patients who were accepted in the EAP but do not receive treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients eligible for the trial are those treated in the EAP of nivolumab in Spain. The total number of patients to be included will be 1400 from 150 participating sites in Spain (anticipated data)
Sampling Method: Non-Probability Sample
Enrollment: 676 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Progression Free survival | At 12 months
  time from inclusion to progression

SECONDARY OUTCOMES:
Overall Response rate | At 12 months
  Percentage of patient reaching a complete, partial or stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Delvys Rodríguez, MD, PhD, Principal Investigator — Hospital Universitario Insular de Gran Canaria; Margarita Majem, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (61):
- Spain (61):
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital de Elche, Elche, Alicante
  - Hospital Universitario de Vinalopó, Elche, Alicante
  - Hospital General Universitario de Elda, Elda, Alicante
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona
  - Hospital de Galdakao, Galdakao, Bizkaia
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Gipuzkoa
  - Centro Oncológico de Galicia, A Coruña, La Coruña
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Universitario Infanta Cristina, Parla, Madrid
  - Hospital Universitario Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital Lluís Alcanyís, Xàtiva, Valencia
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Universitario a Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Vall d' Hebron, Barcelona
  - H. Universitario Quirón Dexeus, Barcelona
  - Hospital de Sant Pau Y de La Santa Creu, Barcelona
  - H. Althaia, Barcelona
  - Hospital Virgen de la Luz, Cuenca
  - Hospital Dr. Josep Trueta, Girona
  - Hospital Clínico San Cecilio, Granada
  - Hospital de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañón, Madrid
  - MD Anderson Cancer Center, Madrid
  - H.U. Puerta de Hierro, Madrid
  - Fundación Jimenez Diaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - H. Carlos Haya, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - H. Morales Messeguer, Murcia
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Son Espases, Palma de Mallorca
  - H. Son Llàtzer, Palma de Mallorca
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital Nuestra Señora Candelaria, Santa Cruz de Tenerife
  - Hospital Virgen del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital General de Valencia, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital de Sagunto, Valencia
  - Hospital La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - H. Miguel Servet, Zaragoza
  - Hospital Universitario de Áraba, Vitoria-Gasteiz, Áraba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.gecp.org